CLINICAL TRIAL: NCT00800670
Title: Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of an Adenovirus-based Tuberculosis Vaccine
Brief Title: Study of the Safety and Immunogenicity of an Adenovirus-based Tuberculosis Vaccine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated after the low dose cohort had been enrolled
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Fiona Smaill, Professor and Chair, McMaster University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB 09-001
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Tuberculosis
Keywords: tuberculosis; vaccine; adenovirus
MeSH Terms: conditions — Tuberculosis; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lower dose (Experimental): Lower dose of Ad5Ag85A: 10^8pfu
  Interventions: Biological: Ad5Ag85A
- Higher dose (Experimental): Higher dose of vaccine Ad5Ag85A: 10^9pfu
  Interventions: Biological: Ad5Ag85A

INTERVENTIONS:
Biological: Ad5Ag85A — Single intra-muscular administration of 10^8 pfu of recombinant-deficient human adenoviral TB vaccine (Ad5Ag85A)
  Arms: Lower dose
Biological: Ad5Ag85A — Single intra-muscular administration of 10^9 recombinant-deficient human adenoviral TB vaccine (Ad5Ag85A)
  Arms: Higher dose

SUMMARY:
The purpose of this Phase 1 study is to evaluate the safety and immune responses of a new tuberculosis vaccine, Ad5Ag85A, administered to healthy volunteers. 48 subjects will be recruited, 24 who have previously been vaccinated with BCG and 24 who have not received BCG vaccine. Two doses of the vaccine will be compared.

DETAILED DESCRIPTION:
As the global tuberculosis (TB) epidemic continues, the incidence of latent and active TB is expected to rise. HIV-infected persons are especially susceptible to TB. An improved TB vaccine over the present BCG vaccine is needed.

The general objectives of our TB vaccine research program are to develop a safe and effective vaccine for persons who at increased risk of contracting TB or reactivating latent tuberculosis and develop a safe booster vaccine for persons who have been previously vaccinated with BCG.

This is an open-labeled phase 1 single institution trial investigating a recombinant genetic TB vaccine AdAg85A given by intramuscular injection in healthy subjects with or without a history of BCG vaccination. Ad5Ag85A is a recombinant replication-deficient adenoviral vector expressing an M. tuberculosis immunogenic antigen Ag85A. We have shown that it is safe, immunogenic and associated with enhanced protection against challenge with virulent M Tb in murine, bovine and guinea pig models. Clinical grade AdAg85A has been manufactured by the Robert E Fitzhenry Vector Laboratory, Centre for Gene Therapeutics, McMaster University, Hamilton, Ontario, Canada.

The effect of pre-existing adenovirus antibodies on the safety and immunogenicity of the recombinant AdTB vaccine will be evaluated and the results of the PPD skin test following vaccination evaluated in a subset of subjects with a history of a negative PPD skin test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human subjects who are between 18 and 55 years of age with or without a history of BCG vaccination.
* HIV antibody negative
* For women, negative pregnancy test and practising two acceptable forms of contraception for the duration of the study (barrier contraceptive, birth control pill, surgically sterile, post-menopausal 2yrs, abstinence)
* For men, using barrier contraception for the duration of the study

Exclusion Criteria:

* Pregnant or lactating women
* Subjects who have any acute or chronic illnesses including active tuberculosis or receiving any drug treatment in the opinion of the investigator likely to affect the immune system.
* Subjects with symptoms suggestive of an upper respiratory tract infection (including cough, runny nose, or sore throat)
* Subjects who have a history of active or latent TB infection or whose PBMCs are strongly responsive to ESAT6/CFP10 stimulation using a commercial interferon gamma release assay for TB [consistent with latent TB infection].
* Subjects who have laboratory values outside the normal range.
* Not available for scheduled follow-up visits. Subjects enrolled in the trial must be followed at 7 days, and then at 2, 4, 8, 16 and 24 weeks post-vaccination.
* Failure to provide written consent.
* Known allergy to vaccine components
* Known exposure to active TB within past 6 months or subjects whose occupation puts them at increased risk of TB exposure (based on Hamilton Health Science/St Joseph Healthcare list of high risk personnel)
* Any abnormality on chest x-ray suggestive of active or remote tuberculosis infection.
* PPD skin test within last 12 months
* BCG status unknown

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Local and systemic signs and symptoms and laboratory toxicity | 24 weeks

SECONDARY OUTCOMES:
Immunogenicity will be compared among the groups by determining the level and quantity of antigen-specific T cells by human interferon ELISA and Elispot assay | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Xing, PhD, Principal Investigator — McMaster University; Fiona M Smaill, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Smaill F, Jeyanathan M, Smieja M, Medina MF, Thanthrige-Don N, Zganiacz A, Yin C, Heriazon A, Damjanovic D, Puri L, Hamid J, Xie F, Foley R, Bramson J, Gauldie J, Xing Z. A human type 5 adenovirus-based tuberculosis vaccine induces robust T cell responses in humans despite preexisting anti-adenovirus immunity. Sci Transl Med. 2013 Oct 2;5(205):205ra134. doi: 10.1126/scitranslmed.3006843. PMID 24089406
- [Result] Jeyanathan M, Damjanovic D, Yao Y, Bramson J, Smaill F, Xing Z. Induction of an Immune-Protective T-Cell Repertoire With Diverse Genetic Coverage by a Novel Viral-Vectored Tuberculosis Vaccine in Humans. J Infect Dis. 2016 Dec 15;214(12):1996-2005. doi: 10.1093/infdis/jiw467. Epub 2016 Oct 4. PMID 27703038